CLINICAL TRIAL: NCT05551104
Title: Safest Choice of Antihypertensive Regimen for Postpartum Hypertension: A Randomized Control Trial (SCARPH)
Brief Title: Safest Choice of Antihypertensive Regimen for Postpartum Hypertension
Acronym: SCARPH
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5220259
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Postpartum Complication; Maternal Hypertension; High Blood Pressure
Keywords: Postpartum Hypertension
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Hypertension | interventions — Nifedipine; Labetalol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Oral Nifedipine (Active Comparator): Participants will receive oral nifedipine for blood pressure control. Dosage may initially start at one 10mg capsule by mouth three times per 24 hours (total of 30mg a day), however dosage may be increased by 30mg increments (i.e. 20mg capsule three times a day for a total of 60mg a day). Maximum dosage for oral Nifedipine will be 120mg per day.
  Interventions: Drug: Oral Nifedipine
- Oral Labetalol (Active Comparator): Participants will receive oral labetalol for blood pressure control. Dosage may initially start at one 200mg tablet by mouth two times per 12 hours (total of 400mg every a day), however dosage may be increased by 100-200mg increments at a time. Maximum dosage for oral labetalol will be 2400mg per day.
  Interventions: Drug: Oral Labetalol

INTERVENTIONS:
Drug: Oral Nifedipine — Administration of oral nifedipine to control postpartum hypertension.
  Other Names: Procardia, Procardia XL
  Arms: Oral Nifedipine
Drug: Oral Labetalol — Administration of oral labetalol to control postpartum hypertension.
  Other Names: Trandate
  Arms: Oral Labetalol

SUMMARY:
The purpose of this investigator-initiated randomized control trial is to determine whether oral Nifedipine versus oral Labetalol is superior in controlling high blood pressures in the postpartum period.

DETAILED DESCRIPTION:
High blood pressure (hypertension) is one of the most common medical disorders in pregnancy and affects 10% of all pregnancies in the United States, with possible short-term and long-term health complications including increased risk of stroke, and liver, kidney, and heart disease. Management of severe high blood pressure after delivery involves medications to lower blood pressure, strict discharge instructions and close follow- up after delivery. Both oral Nifedipine and oral Labetalol are considered safe agents for the treatment of postpartum high blood pressure, however few studies exist that directly compare the two. The investigators want to conduct this study because they want to compare the effects of oral Nifedipine or oral Labetalol on postpartum hypertension. In this study, subjects will get either oral Nifedipine or oral Labetalol. Subjects will not get both. No experimental drugs or devices will be used.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Women who develop postpartum hypertension* after delivery of the placenta or chronic hypertensive postpartum women who require medication for blood pressure control.

  * Postpartum hypertension requiring treatment are defined as systolic blood pressure greater than or equal to 140mmHg or diastolic blood pressure greater than or equal to 90mmHg on at least 2 occasions at least 4 hours apart, or systolic blood pressure greater than or equal to 160mmHg or diastolic blood pressure greater than 110mmHg sustained for more than 15 minutes.

Exclusion Criteria:

* History of moderate persistent asthma, coronary artery disease, heart failure, AV heart block, pulmonary edema
* Contraindication to either Nifedipine or Labetalol
* HR <60 or >110
* Native language other than English or Spanish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Composite maternal morbidity | 0-6 weeks following delivery
  Requiring antihypertensive medication in the postpartum period, readmission for high blood pressure

SECONDARY OUTCOMES:
Length of hospital stay of mothers | Number of hours between time of admission to time of discharge, up to 4 weeks from time of admission.
  The length of hospital stay for mothers will be measured in hours from the time of admission to labor and delivery unit to the time of discharge from the post-partum unit.
Total number of participants who have need for second antihypertensive agent | 0-6 weeks following delivery
  The need to use a second (alternative) antihypertensive medication.

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No